CLINICAL TRIAL: NCT00500786
Title: Safety, Tolerability, Pharmacodynamic Effects and Preliminary Evidence for Efficacy of the Anti-Hypertension Vaccine CYT006-AngQb
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYT006-AngQb 01
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — CYT006-AngQb

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 100 mcg CYT006-AngQb Healthy Volunteers (Experimental)
  Interventions: Biological: CYT006-AngQb
- 100 mcg CYT006-AngQb Hypertensives (Experimental)
  Interventions: Biological: CYT006-AngQb
- 300 mcg CYT006-AngQb Hypertensives (Experimental)
  Interventions: Biological: CYT006-AngQb
- Placebo Healthy Volunteers (Placebo Comparator)
- Placebo Hypertensives (Placebo Comparator)

INTERVENTIONS:
Biological: CYT006-AngQb
  Arms: 100 mcg CYT006-AngQb Healthy Volunteers; 100 mcg CYT006-AngQb Hypertensives; 300 mcg CYT006-AngQb Hypertensives

SUMMARY:
This is a multi-center, randomized, placebo-controlled, time-lagged, parallel-group study in healthy and hypertensive subjects to evaluate safety and tolerability of the vaccine CYT006-AngQb. The trial is double-blind for active vs. placebo within each treatment arm, but open with respect to AngQb dose escalation.

In the first arm, 16 healthy normotensive volunteers are treated with a one dose regimen consisting of a single s.c. injection of 100µg of AngQb or placebo. Upon satisfying safety and tolerability profile, as judged by the independent safety monitoring board, arm two is enrolled.

In arm two 36 patients with mild to moderate hypertension receive three s.c. injections of 100µg CYT006-AngQb (24 patients) or placebo (12 patients). The second and third injections are given 4 and 12 weeks after the first injection, respectively. Upon satisfying safety and tolerability profile, as judged by the independent safety monitoring board, arm three is enrolled.

In arm three 36 patients with mild to moderate hypertension receive three s.c. injections of 300µg CYT006-AngQb (24 patients) or placebo (12 patients). The second and third injections are given 4 and 12 weeks after the first injection, respectively.

The primary objective of the trial is to evaluate safety / tolerability of 3 dose regimens of CYT006-AngQb in healthy volunteers and patients with mild to moderate essential hypertension. Secondary objectives include the assessment of pharmacodynamic effects and their dose-response (immunogenicity and biomarkers of the renin-angiotensin system), and the exploration of clinical efficacy (effects on systolic and diastolic blood pressure)

ELIGIBILITY:
Inclusion Criteria:

* Patients with untreated mild-to-moderate essential hypertension, clinically diagnosed according to the World Health Organization criteria (systolic blood pressure =140-179 mm Hg and/or diastolic blood pressure =90-109 mm Hg on 3 consecutive occasions; standardized after 5 minutes in sitting position)
* Patients with newly diagnosed essential hypertension or previously treated patients from whom antihypertensive therapy can be safely withdrawn for the duration of the study.
* 18 to 65 years of age, males and non-reproductive females (surgically sterilized or post-menopausal)
* Written informed consent
* Patient is willing and able to comply with all trial requirements

Exclusion Criteria:

* Secondary hypertension
* Severe essential hypertension
* Current pharmacological treatment that could affect blood pressure
* Significant renal insufficiency [Serum creatinine > 159 µmol/L (> 1.8 mg/dl)]
* History of cerebrovascular disease
* Type 1 Diabetes or poorly controlled Type 2 Diabetes
* Body mass index (BMI) >32
* Total cholesterol > 6.9 mmol/L (> 266 mg/dl)
* Triglycerides > 3.5 mmol/L ( > 174.3 mg/dl)
* Autoimmune diseases or severe allergies
* Patients with a history of HIV infection, AIDS, hepatitis B or C, or other immunosuppressive disorders
* Current diagnosis or a history of malignancy
* Drug or alcohol abuse within the past 2 years
* Pregnancy or breastfeeding
* Present history of mental diseases
* Participation in any drug trial within three month of onset of current trial
* Previous participation in a clinical trial with a Qb based vaccine (DerQb, NicQb, AllQb)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2004-11; Primary Completion 2006-09 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank D Wagner, MD, Principal Investigator — Parexel International, Berlin, Germany

REFERENCES:
- [Derived] Tissot AC, Maurer P, Nussberger J, Sabat R, Pfister T, Ignatenko S, Volk HD, Stocker H, Muller P, Jennings GT, Wagner F, Bachmann MF. Effect of immunisation against angiotensin II with CYT006-AngQb on ambulatory blood pressure: a double-blind, randomised, placebo-controlled phase IIa study. Lancet. 2008 Mar 8;371(9615):821-7. doi: 10.1016/S0140-6736(08)60381-5. PMID 18328929
- See also: Sponsor's web page — http://www.cytos.com